CLINICAL TRIAL: NCT05053048
Title: A Market Surveillance Study Assessing the Effect of an Alumina Free Device Surface on Bone Mineral Density in Patients Implanted With an SL-PLUS™ Femoral Stem for Total Hip Arthroplasty
Brief Title: Effect of an Alumina Free Device Surface on BMD in Patients Implanted With an SL-PLUS™ Femoral Stem for THA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kantonsspital Baselland Bruderholz (Other)
Collaborators: Smith & Nephew, Inc. (Industry)
Responsible Party: Principal Investigator, Prof. Dr. med. Niklaus F. Friederich, MD, Prof., Kantonsspital Baselland Bruderholz
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20052021
Record Dates: First submitted 2021-08-25; First posted 2021-09-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-08

CONDITIONS: Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Intervention Model Description: Randomised controlles trial, double-blind. Block randomization with block size 10.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- STD-SL-PLUS stem (Experimental): Rectangular SL straight stems made of titanium alloy (Ti-6Al-7Nb). The control stem (STD-SL-PLUS stem) underwent alumina grit blasting to reach the adequate roughness of 4-6 micron.
  Interventions: Device: SL-PLUS-Stem for total hip arthroplasty
- NT-SL-PLUS Stem (Active Comparator): Rectangular SL straight stems made of titanium alloy (Ti-6Al-7Nb). The experimental stem (NT SL-PLUS) underwent alumina grit blasting to reach the adequate roughness of 4-6 micron. The surface of the NT SL-PLUS stem was thereafter additionally treated chemically by short-acid etching with HF and mechanically by dry ice blasting in order to loosen and remove the residual alumina particles up to 96% without changing the existing surface microtopography.
  Interventions: Device: SL-PLUS-Stem for total hip arthroplasty

INTERVENTIONS:
Device: SL-PLUS-Stem for total hip arthroplasty — Patients undergoing primary total hip arthroplasty are randomly assigned (1:1) to receive either an uncemented NT-SL-PLUS Stem (Smith&Nephew Orthopaedics AG, Aarau, Switzerland) or a matching uncemented STD-SL-PLUS stem (Smith&Nephew Orthopaedics AG, Aarau, Switzerland) in a blinded fashion.

SUMMARY:
Alumina particles from the grit blasting of Ti-alloy stems for hip arthroplasty are suspected to contribute to aseptic loosening. An alumina-reduced stem surface was hypothesized to improve osseointegration and show comparable short-term outcomes to those of a standard stem.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older undergoing primary THA for primary or secondary osteoarthritis will be enrolled.

Exclusion Criteria:

* Exclusion criteria were ongoing therapy with cortisone or medications influencing bone metabolism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-08-01 (Actual); Primary Completion 2008-09-30 (Actual); Study Completion 2012-05-31 (Actual)

PRIMARY OUTCOMES:
Baseline Bone mineral density by DEXA | Measurements will be performed 7 days (baseline) after surgery
  Bone mineral density around the stem is measured as a surrogate for prosthesis in-growth by a dual-energy x-ray absorptiometry device (DEXA) (General Electric).
Change from baseline Bone mineral density by DEXA at 3 months | Measurements will be performed 3 months postoperatively
  Bone mineral density around the stem is measured as a surrogate for prosthesis in-growth by a dual-energy x-ray absorptiometry device (DEXA) (General Electric).
Change from baseline Bone mineral density by DEXA at 6 months | Measurements will be performed 6 months postoperatively
  Bone mineral density around the stem is measured as a surrogate for prosthesis in-growth by a dual-energy x-ray absorptiometry device (DEXA) (General Electric).
Change from baseline Bone mineral density by DEXA at 12 months | Measurements will be performed 12 months postoperatively
  Bone mineral density around the stem is measured as a surrogate for prosthesis in-growth by a dual-energy x-ray absorptiometry device (DEXA) (General Electric).
Change from baseline Bone mineral density by DEXA at 24 months | Measurements will be performed 24 months postoperatively
  Bone mineral density around the stem is measured as a surrogate for prosthesis in-growth by a dual-energy x-ray absorptiometry device (DEXA) (General Electric).

SECONDARY OUTCOMES:
Rate of radiolucent lines on hip radiographs (AP and axial) at 12 months | Measurements will be performed at 12 months postoperatively.
  Assessment of radiographs for radiolucent lines (RLs) around the stem.
Rate of radiolucent lines on hip radiographs (AP and axial) at 24 months | Measurements will be performed at 24 months postoperatively.
  Assessment of radiographs for radiolucent lines (RLs) around the stem.
Rate of osteolysis on hip radiographs (AP and axial) at 12 months | Measurements will be performed at 12 months postoperatively.
  Assessment of radiographs for osteolysis around the stem.
Rate of osteolysis on hip radiographs (AP and axial) at 24 months | Measurements will be performed at 24 months postoperatively.
  Assessment of radiographs for osteolysis around the stem.
Rate of hypertrophies and atrophies on hip radiographs (AP and axial) at 12 months | Measurements will be performed at 12 months postoperatively.
  Assessment of radiographs for hypertrophies and atrophies around the stem.
Rate of hypertrophies and atrophies on hip radiographs (AP and axial) at 24 months. | Measurements will be performed at 24 months postoperatively.
  Assessment of radiographs for hypertrophies and atrophies around the stem.
Baseline WOMAC | Measurements will be performed 1 month preoperatively.
  For clinical scoring, the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) will be assessed.
Change in WOMAC at 12 months | Measurements will be performed 12 months postoperatively
  For clinical scoring, the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) will be assessed.
Change in WOMAC at 24 months | Measurements will be performed 24 months postoperatively
  For clinical scoring, the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) will be assessed.
Baseline HHS | Measurements will be performed 1 month preoperatively.
  For clinical scoring, the Harris Hip Score (HHS) will be assessed.
Change in HHS at 12 months | Measurements will be performed 12 months postoperatively
  For clinical scoring, the Harris Hip Score (HHS) will be assessed.
Change in HHS at 24 months | Measurements will be performed 24 months postoperatively
  For clinical scoring, the Harris Hip Score (HHS) will be assessed.
Survival rates | Up to 24 months postoperatively.
  THA survival rates and adverse events will be documented up to 24 months postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Niklaus F. Friederich, MD, Prof., Principal Investigator — Kantonsspital Baselland Bruderholz

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moret CS, Masri SE, Schelker BL, Friederich NF, Hirschmann MT. Unexpected early loosening of rectangular straight femoral Zweymuller stems with an alumina-reduced surface after total hip arthroplasty-a prospective, double-blind, randomized controlled trial. J Orthop Traumatol. 2024 Mar 2;25(1):12. doi: 10.1186/s10195-023-00743-1. PMID 38430413